CLINICAL TRIAL: NCT01721551
Title: Phase 4 Exercise Training in Aspects of Fatigue in Patients Receiving Dialysis Therapy
Brief Title: Sleep and Training Aspects in Dialysis Fatigue - Exercise Intervention
Acronym: StandFirm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Greek Ministry of Development (Other Government); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Research Associate Professor, University of Thessaly
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: UTH2-3/10-10-2012
Record Dates: First submitted 2012-10-26; First posted 2012-11-05 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Fatigue
Keywords: Dialysis fatigue,; exercise intolerance,; muscle atrophy,; cachexia,; disability,; Sleep disorders; Depression; Mental Fatigue,; Cognitive function; Physical Fatigue
MeSH Terms: conditions — Fatigue; Muscular Atrophy; Cachexia; Sleep Wake Disorders; Depression; Mental Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): HD patients will receive a 9 months intradialytic exercise training program
  Interventions: Other: Exercise
- No exercise (Placebo Comparator): HD patients will not participate in any type of systematic exercise training
  Interventions: Other: Usual Treatment

INTERVENTIONS:
Other: Exercise — Training will include a 45-60 min aerobic training on a rehabilitation cycle ergometer (Monark Rehab Trainer 881E) in the supine position during dialysis session. The intensity will progress from 30-40% of the maximum exercise power to 60-70%.
  Arms: Exercise training
Other: Usual Treatment — The CON group received no intervention but the usual treatment
  Arms: No exercise

SUMMARY:
The purpose of the current study is to investigate whether changes in patients' sleep quality and quantity will be followed by improvements in parameters related to physical and mental fatigue in patients receiving hemodialysis therapy.

More specific, the current project will investigate the effect of a 9 months intradialytic exercise training in aspects related to fatigue, quality of life and depression.

DETAILED DESCRIPTION:
Chronic renal disease is a "silent epidemic" affecting up to 10% of the population in the EU, USA, and Asian with some of the sufferers progressing into end-stage renal failure.

Renal disease patients are characterized by progressively worsening muscle weakness and muscle atrophy due to both a metabolic and a disuse component collectively described as uremic myopathy. While various interventions in stable HD patients have helped these patients improve their functionality, they still have not proven enough to bring their muscle quality and quantity up to the levels of a healthy sedentary person. Moreover, patients present with sleep problems, neurological and quality of life issues, anxiety and/or symptoms of depression but most notably they complain of chronic fatigue and "lack of energy".

Other factors that contribute to the excessive fatigue are a lack of restorative sleep, excess pre-dialysis weight, poor nutritional status, restless legs syndrome and the overall mental status of the patients. Evidently, of all of these factors can contribute to a self-exacerbating process, a vicious circle, of fatigue due to inactivity and further inactivity due to fatigue. This sensation of an enduring fatigue interferes with physical and social activities and feeds perceptions of increased restrictions and barriers, and leads to a significant reduction of physical activity and functional capacity, which in turn contributes to the increased cardiovascular risk and a high mortality rate among these patients.

Rationale: The investigators hypothesize that by improving the patients fitness levels, it will lead in more energy during day and therefore less fatigue. Our mission is to help the HD patient to better cope with their sensation of fatigue.

ELIGIBILITY:
Inclusion Criteria:

Adult hemodialysis patients both sexes who has received regular HD treatment for at least 6 months, adequate dialysis delivery with Kt/V >1.1 and good compliance with dialysis treatment, with serum albumin > 2.5 g/dL, hemoglobin>= 11g/dL sleep onset latency > 15 minutes or sleep efficiency < 85% or arousal index > 25

Exclusion Criteria:

Patients unable to give informed consent, with opportunistic infection in the last 3 months, malignancy or infection requiring intravenous antibiotics within 2 months prior to enrollment, myoskeletal contraindication to exercise requirement for systemic anticoagulation, participating or participated in an investigational drug or medical device study within 30 days or five half-lives, pregnant, breast feed or female of childbearing potential who does not agree to remain abstinent or to use an acceptable contraceptive regimen, lactate dehydrogenase > 300U/L, prolonged heart wave (QT) interval (as defined by corrected QT (QTc) > 460 msec in males and > 470 msec in females) on screening electrocardiogram (ECG), known current alcohol or drug abuse, known or suspected hypersensitivity to the study medication or any of its ingredients,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Levels of Fatigue | 9 months
  Fatigue will be assessed by direct and indirect measurements. Physical Fatigue will be assessed by hand grip, functional tests, cardiorespiratory max test. Mental Fatigue will be assessed by questionnaires. Cognitive Fatigue will be assessed by questionnaires. Pre and Post dialysis fatigue will be assessed by hand grip and questionnaires.

SECONDARY OUTCOMES:
Body composition | 9 months
  Muscle composition will be assessed by BCM bio impedance system
Muscle Functionality | 9 months
  Muscle functionality will be assessed by functional tests. Muscle Fatigue will be assessed by a fatigue protocol.

OTHER OUTCOMES:
Quality of life aspects | 9 months
  Depression, Quality of life will be assessed by questionnaires. Sleep quality and quantity will be assessed by questionnaires and a full night polysomnography.
Cardiac functionality | 9 months
  Structural and functional characteristics of the heart will be assessed by an ecocardiography system before, during and after hemodialysis
Neurological Assessment | 9 months
  Full neurological assessment will take place

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos K. Sakkas, PhD, Principal Investigator — Center for Research and Technology Thessaly - University of Thessaly; Christina Karatzaferi, PhD, Principal Investigator — University of Thessaly; Ioannis Stefanidis, MD, PhD, Study Director — University of Thessaly
Locations (3):
- Greece (3):
  - University Hospital of Larissa, Larissa, Thessaly
  - Patsidis General Clinic, Larissa, Thessaly
  - General Hospital of Trikala, Trikala, Thessaly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakkas GK, Karatzaferi C. Hemodialysis fatigue: just "simple" fatigue or a syndrome on its own right? Front Physiol. 2012 Jul 31;3:306. doi: 10.3389/fphys.2012.00306. eCollection 2012. No abstract available. PMID 22934057
- [Background] Grigoriou SS, Giannaki CD, George K, Karatzaferi C, Zigoulis P, Eleftheriadis T, Stefanidis I, Sakkas GK. A single bout of hybrid intradialytic exercise did not affect left-ventricular function in exercise-naive dialysis patients: a randomized, cross-over trial. Int Urol Nephrol. 2022 Jan;54(1):201-208. doi: 10.1007/s11255-021-02910-x. Epub 2021 Jun 7. PMID 34100215
- [Background] Grigoriou SS, Krase AA, Karatzaferi C, Giannaki CD, Lavdas E, Mitrou GI, Bloxham S, Stefanidis I, Sakkas GK. Long-term intradialytic hybrid exercise training on fatigue symptoms in patients receiving hemodialysis therapy. Int Urol Nephrol. 2021 Apr;53(4):771-784. doi: 10.1007/s11255-020-02711-8. Epub 2021 Jan 2. PMID 33387217
- [Background] Grigoriou SS, Karatzaferi C, Sakkas GK. Pharmacological and Non-pharmacological Treatment Options for Depression and Depressive Symptoms in Hemodialysis Patients. Health Psychol Res. 2015 Apr 13;3(1):1811. doi: 10.4081/hpr.2015.1811. eCollection 2015 Apr 13. PMID 26973957
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639